CLINICAL TRIAL: NCT01194869
Title: Phase II Neoadjuvant Trial of Sorafenib in Combination With Cisplatin Followed by Dose Dense Paclitaxel for ER-, PR-, Her2- (Triple Negative) Early-Stage Breast Cancer
Brief Title: Preoperative Trial of Sorafenib in Combination With Cisplatin Followed by Paclitaxel for Early Stage Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual, availability of other clinical options
Sponsor: Emory University (Other)
Collaborators: Amgen (Industry); Bayer (Industry)
Responsible Party: Principal Investigator, Elisavet Paplomata, MD, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00019781; WCI1590-08 (Other: Other)
Record Dates: First submitted 2010-09-01; First posted 2010-09-03 (Estimated); Results first posted 2016-07-28 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Sorafenib; Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib (Experimental): Sorafenib 400 mg twice daily throughout the study. Patients will receive this as a single-agent for the first four weeks, then in combination with cisplatin followed by paclitaxel.
  Interventions: Drug: Sorafenib; Drug: Cisplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Sorafenib — Sorafenib 400 mg twice daily throughout the study. Patients will receive this as a single-agent for the first four weeks, then in combination with cisplatin followed by paclitaxel.
  Other Names: Nexavar
Drug: Cisplatin — 75 mg/m² given IV
  Other Names: Platinol; CDDP; Cis-diamminedichloroplatinum(II)
Drug: Paclitaxel — 175 mg/m² given IV
  Other Names: Taxol

SUMMARY:
The purpose of this study is to identify new treatment regimens with better response rates and to find out if the combination of cisplatin and sorafenib followed by paclitaxel and sorafenib can shrink the size of your breast tumor and allow you to preserve your breast. Sorafenib is a newer drug that targets blood vessel formation and may help the chemotherapy work better. Additionally, by receiving chemotherapy before surgery, we will be able to determine if your cancer is responsive to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive breast carcinoma.
* Early stage breast cancer (Stage I (tumor size ≥ 1cm), II and IIIA).
* Invasive breast cancer must be estrogen receptor (ER)-negative, progesterone receptor (PR)-negative, human epidermal growth factor receptor 2 (Her2)-negative. If breast cancer is Her2 2+ by immunohistochemistry (IHC), then fluorescence in situ hybridization (FISH) must be negative for Her2 gene amplification.
* No evidence of disease outside the breast or chest wall, except ipsilateral axillary lymph nodes.
* Patients must have measurable disease as defined by palpable lesion with both diameters ≥ 1cm measurable with caliper and/or a positive mammogram or ultrasound with at least one dimension ≥ 1cm. Screening mammogram of the contralateral breast must be performed within past 12 months per standard practice guidelines. Clip placement is required for study entry. Baseline measurements of the indicator lesions must be recorded on the Patient Registration Form. To be valid for baseline, the measurements on clinical exam must have been made within 14 days if the mass is palpable. If the mass is not palpable, a mammogram or MRI must be done within 14 days. If the mass is palpable, a diagnostic mammogram of the affected breast or MRI must be done within 2 months prior to study entry.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 within 14 days of study entry.
* Normal (greater than 50%) left ventricular ejection fraction (LVEF) by multigated acquisition (MUGA) scan or echocardiography.
* Signed informed consent.
* Adequate organ function within 2 weeks of study entry:

  * Absolute neutrophil count ≥ 1000/mm³, Hgb ≥ 9.0 g/dl and platelet count ≥ 100,000/mm³
  * Total bilirubin ≤ upper limit of normal
  * Creatinine ≤ 1.5 mg/dL or calculated creatinine clearance (CrCL) ≥ 50 mL/min using the Cockroft Gault equation
  * Serum glutamic oxaloacetic transaminase (SGOT)(AST) or serum glutamic pyruvic transaminase (SGPT)(ALT) and alkaline phosphatase must be within the range allowing for eligibility
* Patients must be ≥ 18 years.
* International normalized ratio (INR) < 1.5 or a prothrombin time (PT)/partial thromboplastin time (PTT) within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment.
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation.
* Patients with history of breast cancer greater than 5 years from initial diagnosis and are disease free are eligible for the study. Patients with history of ductal carcinoma in situ (DCIS) are eligible if there were treated with surgery alone.

Exclusion Criteria:

* Prior chemotherapy, hormonal therapy, biologic therapy, investigational agent, targeted therapy or radiation therapy for current breast cancer.
* Metastatic disease on baseline staging scans.
* Medical, psychological or surgical condition which the investigator feels might compromise study participation.
* History of previous or current malignancy at other sites with the exception of adequately treated carcinoma in-situ of the cervix or basal or squamous cell carcinoma of the skin. Patients with a history of other malignancies, who remain disease free for greater than five years are eligible.
* Evidence of grade 2 or greater sensory and/or peripheral neuropathy.
* Serious, uncontrolled, concurrent infection(s).
* Major surgery within 4 weeks of the start of study treatment, without complete recovery.
* Pregnant or lactating women are not eligible. Women or men of childbearing potential not using a reliable and appropriate contraceptive method are not eligible. (Postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential).
* Use of St. John's Wort or rifampin (rifampicin).
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.
* Any condition that impairs patient's ability to swallow whole pills.
* Any malabsorption problem.
* Evidence or history of bleeding diathesis or coagulopathy.
* Known human immunodeficiency virus (HIV) infection or chronic hepatitis B or C.
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Pulmonary hemorrhage/bleeding event ≥ Common Toxicity Criteria for Adverse Effects (CTCAE) Grade 2 within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event ≥ CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Cardiac disease: congestive heart failure > class II New York Heart Association (NYHA). Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Known brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisavet Paplomata, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at Winship Cancer Institute of Emory University, Emory University Hospital Midtown, and Grady Health System. The study closed to accrual in June 2015.
Period: Overall Study
Arm/Group | Sorafenib
Started | 25
Completed | 21
Not Completed | 4
Not completed — Disease Progression | 2
Not completed — Toxicity | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 42 [34 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR) at the Time of Surgery After Preoperative Treatment
Description: Pathologic complete response (pCR): Absence of invasive breast cancer in the breast (mastectomy or lumpectomy) specimen at the time of definitive surgery. Presence of in situ cancer alone will be considered a pCR but may be recorded separately.
Time Frame: At the time of surgery, after 24 weeks of preoperative treatment
Measure: Number; unit: participants
Arm/Group | Sorafenib
Number analyzed (Participants) | 21
participants | 5

2. Secondary Outcome: Clinical Response Rate During Follow-up (Disease Recurrence)
Description: Response will be assessed according to World Health Organization criteria with progressive disease (PD) defined as a 25% or greater increase in a single lesion, OR reappearance of any lesion which has disappeared, OR clear worsening of any evaluable disease OR appearance of any new lesion/site.
Time Frame: Up to 2 years after definitive surgery
Measure: Number; unit: participants
Arm/Group | Sorafenib
Number analyzed (Participants) | 21
participants | 6

3. Secondary Outcome: Clinical Response Rate (Complete Pathologic Response Rate After Surgery)
Description: Pathologic complete response (pCR): Absence of invasive breast cancer in the breast (mastectomy or lumpectomy) specimen during follow-up. Presence of in situ cancer alone will be considered a pCR but may be recorded separately.
Time Frame: Up to 2 years after definitive surgery
Measure: Number; unit: participants
Arm/Group | Sorafenib
Number analyzed (Participants) | 21
participants | 0

ADVERSE EVENTS:
Arm/Group | Sorafenib
Serious Adverse Events (participants affected / at risk) | 6/25
Other Adverse Events (participants affected / at risk) | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=25)
Obstructive Jaundice (Hepatobiliary disorders) | 1
Acute Stroke (Nervous system disorders) | 1
Pulmonary Embolus (Vascular disorders) | 1
Death (General disorders) | 2
Chest Pain (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=25)
Fatigue (General disorders) | 19
Hand-Foot Syndrome (General disorders) | 13
Hypertension (Vascular disorders) | 11
Neuropathy (Nervous system disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes